CLINICAL TRIAL: NCT06197906
Title: Effectiveness and Safety of the RIGHTEST™ Continuous Glucose Monitoring System for Blood Glucose Management in Persons With Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bionime Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CN-312-01
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DM self-control group (Other)
  Interventions: Device: Device implant

INTERVENTIONS:
Device: Device implant — subcutaneous device implanting

SUMMARY:
The trial is expected to enroll 120 confirmed cases of type 1 or type 2 diabetes. All eligible subjects must wear a continuous glucose monitoring system on both the left and right upper arms for a maximum of 15 days (360 hours) and adhere to the clinical visit protocol. The entire trial process consists of pre-screening visits, 5 clinical visits, and 1 telephone follow-up.

After enrollment, all subjects will be randomly assigned to either Group A or Group B to determine the time points for clinical visits. Group A subjects will have venous blood drawn on days 1 and 10 (±1) post-wearing, while Group B subjects will have venous blood drawn on days 5 (±1) and 15 (-1) post-wearing. All subjects will remove all devices on day 15 (-1) based on system prompts and undergo a telephone follow-up on day 4 (±3) thereafter. This clinical trial does not involve long-term follow-up.

During the trial, the blood glucose values measured by the "continuous glucose monitoring system" worn by the subjects will be analyzed against the EKF venous blood glucose values measured at the medical institution on days 1, 5 (±1), 10 (±1), and 15 (-1) as control reference values. This analysis aims to evaluate the accuracy, repeatability, stability, high and low blood glucose event alerts, and safety of the continuous glucose monitoring system.

Additionally, fingertip blood glucose measurements taken by subjects during home use will be collected to assess the operational feasibility of the continuous glucose monitoring system in a home setting.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are aged 18 to 80 years old.
2. Participants have been diagnosed with type 1 or type 2 diabetes.
3. Participants must meet one of the following treatment criteria:

   * Daily insulin injections and/or insulin pump therapy at least once a day.
   * Use of antidiabetic medications, with glycated hemoglobin (HbA1c) not less than 8%. Relevant medications include but are not limited to: sulfonylureas, biguanides, α-glucosidase inhibitors, thiazolidinediones, dipeptidyl peptidase 4 inhibitors, sodium-glucose cotransporter-2 inhibitors, and glucagon-like peptide 1 receptor agonists (GLP-1RAs).
4. Participants who can comply with the experimental procedures and related requirements specified in the protocol.
5. Volunteers willing to participate in this trial and who have signed the informed consent form.

Exclusion Criteria:

1. Known allergy to disinfectant alcohol or medical-grade skin patches.
2. Presence of skin trauma, infection, or skin disease at the site where the trial device is to be worn.
3. Hemoglobin levels less than 90.0g/L.
4. Estimated glomerular filtration rate (eGFR) less than 30 mL/min/1.73m2.
5. Use of other implanted medical devices, such as pacemakers or defibrillators.
6. Acutely critically ill patients.
7. Patients with active infectious diseases.
8. Requirement for imaging examinations, phototherapy, or thermotherapy during the wearing period.
9. History of unconscious hypoglycemia in the six months preceding the trial; patients admitted to the hospital at screening are excluded.
10. Pregnant women or women planning to become pregnant during the study.
11. Inability to read the product instructions or inability to wear the trial device after receiving education and training.
12. Participation in another clinical trial within the two weeks prior to screening.
13. Other situations determined by the investigator as unsuitable for participation in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
accuracy | 15 day
  The percentage of the CGM System raw readings within ±20/20%of paired reference measurements across the device measuring range overall are evaluated.